CLINICAL TRIAL: NCT02754648
Title: Three Different Laparoscopic Approaches for Ovarian Endometrioma and the Effect on Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Assistant professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ain ShamsU Laparoscopic Unit
Record Dates: First submitted 2016-03-16; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A; laparoscopic ovarian endometrial aspiration (Active Comparator): Laparoscopic ovarian endometrial aspiration will be done for thirty patients with ovarian endometriotic cyst. .
  Interventions: Procedure: laparoscopic ovarian endometriotic cyst
- group B; laparoscopic ovarian endometrial stripping (Active Comparator): Laparoscopic ovarian endometrial stripping will be done for thirty patients with ovarian endometriotic cyst.
  Interventions: Procedure: laparoscopic ovarian endometriotic cyst
- Group c laparoscopic ovarian endometrial de-roofing (Active Comparator): Laparoscopic ovarian endometrial de-roofing and bed cauterization will be done for thirty patients with ovarian endometriotic cyst.
  Interventions: Procedure: laparoscopic ovarian endometriotic cyst

INTERVENTIONS:
Procedure: laparoscopic ovarian endometriotic cyst

SUMMARY:
Is ovarian reserve and fecundity rate higher with laparoscopic ovarian aspiration rather than laparoscopic ovarian cystectomy and laparoscopic ovarian de-roofing in infertile woman with ovarian endometrioma or not?

DETAILED DESCRIPTION:
Primary objective:

To assess antral follicular count before and after treatment of endometriotic cyst either by aspiration, stripping, de-roofing and bed cauterization.

Secondary objectives To assess anti mullerian hormone level, follicle stimulating hormone level ,Doppler blood flow before and after treatment of endometriotic cyst either by aspiration, stripping, de-roofing and bed cauterization.

ELIGIBILITY:
Inclusion Criteria:

* Infertile woman aged 18-35 years old.
* Endometriotic ovarian cyst with size less than or equal 5 cm.

Exclusion Criteria:

* Other than included criteria.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The antral follicular count which records the number of visible ovarian follicle (2-10 mm mean diameter) seen by transvaginal ultrasound on menstrual cycle( days 2_5) | One month
  Cut point(3-10)

SECONDARY OUTCOMES:
Anti mullerian hormone level in blood secreted by antral follicles 2-6 mm diameter in ovary | One month
  Measure in ng/ml cut point is( 0.2-0.7)
Follicle stimulating hormone in blood secreted by antral follicles on day 2-4 of menstrual cycle | One month
  Cut point is(10-20) measured in international unit/litre

IPD SHARING:
Plan to Share IPD: No